CLINICAL TRIAL: NCT06438978
Title: An Open-Labelled, Phase I Clinical Trial to Assess the Safety Reactogenicity, Tolerability and Immunogenicity of a Tuberculosis Vaccine BBV169 (MTBVAC), in Healthy Indian Adults
Brief Title: Tuberculosis Vaccine in Healthy Indian Adults
Acronym: BBV169/2023
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bharat Biotech International Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: BBIL/MTBVAC/2023; BBIL/MTBVAC/2023 (Other: Bharat Biotech International Limited)
Record Dates: First submitted 2023-12-11; First posted 2024-06-03 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis | interventions — Tuberculosis Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MTBVAC (Experimental): 30 healthy, BCG vaccinated, HIV negative, adults, aged 18 - 65 years, in whom LTB Infection has been excluded by negative QuantiFERON® (QFT) Gold-Plus assay.
  Interventions: Biological: Tuberculosis Vaccine

INTERVENTIONS:
Biological: Tuberculosis Vaccine — 1. Live, attenuated Mycobacterium tuberculosis (M. tb)- MTBVAC (MTBVAC)01 strain
  2. 3-17x105CFU (Per dose) Sucrose Sodium glutamate
  3. Lyophilized pellet in vials (10doses)
  4. 0.1 mL/dose (After reconstitution with 1 mL/vial sterilized water for injection)

SUMMARY:
An Open-labelled, Phase I Clinical Trial to Assess the Safety, Reactogenicity, Tolerability, and Immunogenicity of MTBVAC in healthy Indian adult volunteers A total of 30 subjects with Quantiferon®-TB Gold Plus assay negative and ages 18 to 65 years will be enrolled in this trial. All the subjects will receive a single dose of MTBVAC via the intradermal route in the right deltoid region. DSMB meetings will be conducted after Day 28 , Day 90 & Day 180 after vaccinating all subjects.

DETAILED DESCRIPTION:
An Open-labelled, Phase I Clinical Trial to Assess the Safety, Reactogenicity, Tolerability, and Immunogenicity of MTBVAC in healthy Indian adult volunteers A total of 30 subjects with Quantiferon®-TB Gold Plus assay negative and ages 18 to 65 years will be enrolled in this trial. All the subjects will receive a single dose of MTBVAC via the intradermal route in the right deltoid region. DSMB meetings will be conducted after Day 28 , Day 90 & Day 180 after vaccinating all subjects.

Study Objectives:

Primary Objective To evaluate the safety and reactogenicity of MTBVAC

End points:

1. The occurrence of immediate adverse events within 30mins of vaccination [Time Frame: 30 mins].
2. The occurrence of solicited adverse events within fourteen days of vaccination [Time Frame: daily follow- up for 14 days].
3. The injection site reactions will be followed-up for 90 days.
4. The occurrence of any unsolicited adverse events throughout the study duration [Time Frame: throughout the trial duration].
5. The occurrence of serious adverse events (SAEs) [Time Frame: throughout the trial duration].
6. AESI (Adverse Event of Special Interest) is to be considered throughout the trial period.
7. Hematological, biochemical safety test levels before and after vaccination

Study design:

An Open-labelled, Phase I Clinical Trial to Assess the Safety, Reactogenicity, Tolerability, and Immunogenicity of MTBVAC in healthy Indian adult volunteers A total of 30 subjects with Quantiferon-TB Gold Plus assay negative and ages 18 to 65 years will be enrolled in this trial. All the subjects will receive a single dose of MTBVAC via the intradermal route in the right deltoid region. DSMB meetings will be conducted after Day 28 , Day 90 & Day 180 after vaccinating all subjects

1. Safety Lab investigations -10ml of blood on Day of screening, Day 28, 90,180.
2. Sputum GeneXpert Ultra Test - Sputum sample at screening for all participants and participants with suspected TB
3. Urine test- CUE for all participants at screening, Day 28,90,180 and UPT (female participant of the child bearing age group) on Day0 ,28,90,180
4. Quantiferon Gold Plus assay -5ml of blood on Day of screening, Day 28,90 ,180.
5. Antigen specific CD4/CD8 response--10ml of blood atDay0, 28,90 180.

Study Procedure:

Visit1: Screening-7 to 0

1. Screening of healthy adults of age 18-65 years to assess eligibility by inclusion and exclusion criteria for the trial will take place.
2. After obtaining written informed consent from the healthy participants,
3. Demographic information (age, gender, date of birth, weight [kg], and height [cm], body mass index, address(corresponding and permanent), Contact number, alcohol consumption/substance use, and smoking status/tobacco use),medical history, co-morbid conditions and concomitant medication will be noted,
4. A physical examination of the subject will be carried out. ECG, Chest X-ray, USG abdomen, and sputum for AFB & GeneXpert ultra test will be done for all subjects.
5. 10ml of the blood sample will be collected for screening lab investigations which include CBP, liver function tests, kidney function tests, lipid profile, ESR, RBS, CRP, CUE, TSH, beta HCG (female subjects of, child bearing age group), and serology for HIV1 and 2, HbsAg and HCV.
6. 5ml of the blood sample will be collected for Quantiferon Gold Plus assay.
7. QFT Plus negative subjects will be recruited.

Visit 2:Baseline Day 0

1. From the eligible subjects (in good general health or stable preexisting disease as per the discretion of the principal investigator), blood samples will be withdrawn for Immunogenicity analysis, and urine for UPT [for females of child bearing potential] will be done before vaccination.
2. After administration of the trial vaccine, the subjects will remain at the trial site for at least 30 minutes of observation to record any immediate adverse event.
3. An injection site Photograph will be captured after the assessment of injection site reactions.
4. Diary cards will be distributed to the subjects.
5. Telephonic follow-up is done for 6 days to assess the solicited events and health status.

Visit3: Day7+1

1. The subjects will visit the trial site 7 days after vaccination for safety assessment, which includes solicited and unsolicited adverse events, medical history, vital signs, physical examination, and concomitant medications. The participant will be interviewed for any suspected TB symptoms and concomitant medication. During this visit, the trial personnel will review and collect the diary card.
2. New Diary card will be distributed.
3. An injection site photograph will be captured after the assessment of injection site reactions.
4. Telephonic follow-up will be done for next 7 days to assess the solicited events and health status

Visit4: Day 28±2

1. The subjects will visit the trial site 28±2 days after vaccination. During this visit, the subjects will be examined physically and the history of any adverse events, suspected TB symptoms, and concomitant medications will be asked. The trial personnel will review and collect the diary card. Blood samples will be withdrawn to assess Immunogenicity and safety lab investigations-CBP, Liver function tests, Kidney function tests, Lipid Profile, ESR, CRP and RBS.
2. An injection site photograph will be captured after assessment of injection site reactions
3. Urine samples will be collected for complete urine examination for all and UPT [wherever required]

Visit5: Day 90+7

1. The subjects will visit the trial site 90+7 days after vaccination. During these visits, the subjects will be physically examined and a history of any adverse events, suspected TB symptoms and concomitant medications will be asked. Injection site Photograph will be captured after assessment of injection site reactions. Blood samples will be withdrawn to assess Immunogenicity and safety lab investigations- CBP, Liver function tests, Kidney function tests, Lipid Profile, ESR, CRP and RBS.
2. Urine samples will be collected for complete urine examination for all and UPT [wherever required]

Visit6:Day180+7

1. The subjects will visit the trial site 6 months after vaccination. During this visit, the subjects will be physically examined and the history of any adverse events suspected TB symptoms, and concomitant medications will be asked. Injection site Photograph will be captured after assessment of injection site reactions. Blood samples will be withdrawn to assess Immunogenicity and safety lab investigations-CBP, Liver function tests, Kidney function tests, Lipid Profile, ESR, CRP and RBS
2. Urine samples will be collected for complete urine examination for all and UPT [wherever required]

Visit for Clinically suspected TB during follow-up:

1. If any participant develops TB symptoms (including but not limited to persistent cough, hemoptysis, fever, unintended weight loss, fatigue or lethargy, night sweats, or pleuritic chest pain) during the follow-up after vaccination, he/she will be advised to report to the trial clinic.
2. A detailed medical history with a thorough physical examination will be done.

Based on the results subjects will be classified as follows:

1. In suspected PTB, the trial investigator will undertake investigations (bacteriological, microbiological, and radiological) as per National Tuberculosis Elimination Program (NTEP) guidelines for confirming PTB. If confirmed, the trial investigator will provide/refer participant to concerned department for the required treatment as per NTEP guidelines and will ensure safety follow-up till the end of the trial.
2. In suspected EPTB, the trial investigator will undertake the required investigations for confirming the diagnosis of EPTB as per NTEP guidelines. If confirmed, the trial investigator will provide/refer participant to concerned department for the required treatment as per NTEP guidelines and will ensure safety followup till the end of the trial.
3. If any subject is confirmed with any form of TB, they will not be assessed for Immunogenicity further, But safety will be followed up to 180days
4. If the participant is not diagnosed with TB (PTB or EPTB) as per NTEP guidelines, he/she will be continued in to the trial and followed up till the end of the trial period.
5. All the TB cases will be reviewed by the Adjudication committee

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide written informed consent.[Audio video consent for vulnerable subjects]
2. Participants of either gender of age between ≥18 to ≤65years.
3. Only QFT negative participants will be included
4. Good general health as determined by the discretion of the investigator (vital signs (heart rate ≥60 to≤100 bpm; blood pressure systolic ≥90 mm Hg and <140 mm Hg; diastolic ≥ 60 mm Hg and <90 mm Hg; oral temperature <100.4ºF), medical history, and physical examination).
5. Expressed interest and availability to fulfill the study requirements.
6. For a female participant of childbearing potential, planning to avoid pregnancy (use of an effective method of contraception or abstinence) from the time of study enrolment until at least 3 months after IP administration.
7. Male subjects of reproductive potential: Use of condoms to ensure effective contraception with the female partner from IP administration until 3 months.
8. No evidence of active TB disease during screening - Normal chest radiograph and no bacteriological positivity by Genexpert plus test of sputum for M. tb
9. Clinically acceptable laboratory values for blood tests and a negative pregnancy test (for childbearing-age women)
10. Seronegative for human immunodeficiency virus 1 and -2 (HIV- 1/2) antibodies, hepatitis B surface antigen (HBsAg), and hepatitis C virus (HCV) antibodies.
11. Had BCG vaccination at Birth, documented through medical history or presence of scar.

    -

Exclusion Criteria:

1. Any chronic febrile illness with oral temperature > 100°F on the day of enrollment.
2. Evidence of pulmonary pathology as confirmed by chest X-ray.
3. History of any form of TB Disease.
4. Prior or present anti-TB treatment
5. Received Tuberculin Skin Test (TST) within 3 months (90 days) prior to Study Day 0.
6. Clinical evidence of Active TB
7. Subjects with house hold contacts of Active TB
8. History of allergic reactions (significant IgE-mediated events) or anaphylaxis to previous immunizations (any vaccine).
9. QFT Plus positive subjects.
10. History of allergic disease or reactions.
11. History of previous administration of experimental Mycobacterium tuberculosis vaccines.
12. Use of any investigational or non-registered product (drug or vaccine) in another experimental protocol other than the trial vaccines within 30 days preceding the vaccination, or planned use during the trial period.
13. Any chronic drug therapy to be continued during the trial period.
14. Chronic administration of immune suppressors or other immune- modifying drugs.
15. Administration of any immunoglobulins, any immunotherapy, and/or any blood products within the three months preceding the vaccination, or planned administrations during the trial period.
16. Any confirmed or suspected immunosuppressive or immunodeficient condition (including HIV) based on medical history and physical examination.
17. Any condition or history of any acute or chronic illness or medication, which, in the opinion of the Investigator, may interfere with the evaluation of the trial objectives.
18. A family history of congenital or hereditary immunodeficiency.
19. History of any neurologic disorders or seizures.
20. History of chronic alcohol consumption and/or drug abuse.
21. Major congenital defects.
22. Pregnant or lactating female.
23. Female planning to become pregnant or planning to discontinue contraceptive precautions until 3 months.
24. Those who have been vaccinated with live attenuated vaccines within 30 days of trial vaccine administration and those who are planning to take live attenuated vaccine within 30 days after trial vaccine administration 25 . Administration of any vaccines that are not live attenuated 30 Days before trial vaccine administration -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-01-19 (Actual); Primary Completion 2024-01-29 (Actual); Study Completion 2024-07-27 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and reactogenicity of MTBVAC Immediate reaction | 30 Minutes of vaccination.
  Adverse reactions after administration of each dose
To evaluate the safety and reactogenicity of MTBVAC-Solicited adverse events | 14 days
  Incidence, intensity, and the causality of all solicited adverse events during the 14-day follow up period after each dose.
To evaluate the safety and reactogenicity of MTBVAC-injection site reactions | 90 Days
  The injection site reactions will be followed-up for 90days.
To evaluate the safety and reactogenicity of MTBVAC-unsolicited adverse events | Through out the trial duration till Day180 Days
  The occurrence of any unsolicited adverse events throughout the study duration
To evaluate the safety and reactogenicity of MTBVAC-Serious Adverse Events (SAEs) | Through out the trial duration till Day180 Days
  Incidence, intensity, and the causality of all adverse events and Serious Adverse Events (SAEs) during the entire study period.
To evaluate the safety and reactogenicity of MTBVAC-AESI (Adverse Event of Special Interest) | Through out the trial period till Day180 Days
  AESI (Adverse Event of Special Interest) is to be considered throughout the trial period.
To evaluate the safety and reactogenicity of MTBVAC-Hematological safety test levels before and after vaccination | before and after vaccination on Day 0
  Hematological safety test levels before and after vaccination
To evaluate the safety and reactogenicity of MTBVAC-Biochemical safety test levels before and after vaccination | before and after vaccination on Day 0
  Biochemical safety test levels before and after vaccination

SECONDARY OUTCOMES:
Cellular immune responses | Days 28
  Cellular immune responses [QFT Plus ] at Days 28
Cellular immune responses | Days 90
  Cellular immune responses [QFT Plus ] at Days 90
Cellular immune responses | Days 180
  Cellular immune responses [QFT Plus ] at Days 180.
Antigen-specificCD4/CD8 response | Days 0,28,90 and 180
  Antigen-specificCD4/CD8responseatDays0, 28, 90 and 180

CONTACTS AND LOCATIONS:
Overall Officials: Dr.V.Krishna Mohan, PhD, Study Director — Bharat Biotech International Limited
Locations (1):
- NIMS, Hyderabad, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: No